CLINICAL TRIAL: NCT05213403
Title: Innovative "Scoring System" in Breast Cancer: a Valid Surgical Choice After Neoadjuvant Chemotherapy
Brief Title: Innovative "Scoring System" in Breast Cancer Post Neoadiuvant Chemotherapy
Acronym: BreastNESSy
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FABI ALESSANDRA, Dr.ssa, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4694
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient G1: Correlation between surgery and scoring system
  Interventions: Diagnostic Test: Evaluation with new scoring system
- Patients G2: Incongruence between surgery and scoring system
  Interventions: Diagnostic Test: Evaluation with new scoring system

INTERVENTIONS:
Diagnostic Test: Evaluation with new scoring system — Evaluate whether patients who have received surgery in line with the developed "scoring system" have a better aesthetic and oncological outcomes

SUMMARY:
Our aim is to create a Scoring System (SS) able of guaranteeing radical oncology by completely removing cancer and aesthetic outcomes in line with the needs or expectations of the patients that helps surgeons to decide the type of surgery in patients undergoing NACT.

Secondary outcome is to assess the ability of the score to avoid neoplastic relapses by evaluating:

* Loco-regional disease free-survival (LR-DFS): months between start of NACT and date of a neoplastic recurrence in residual mammary gland, in ipsilateral chest wall or in ipsilateral axilla.
* Distant disease-free survival (DDFS): months between start of NACT and date of onset of visceral or skeletal metastases.
* Overall survival (OS): months from the start of NACT to death or last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing neoadjuvant chemotherapy
* Surgery: Breast conservative surgery; Oncoplastic surgery type II; Conservative mastactomy (nipple sparing - NSM or skin sparing - SSM)

Exclusion Criteria:

* lack of initial staging or restaging;
* previous or synchronous history of systemic malignant neoplasms.
* history of homo-or contralateral breast cancer.
* initial evidence of metastatic pathology or development of metastases during noeadjuvant chemotherapy (Stage IV)
* indication to modified radical mastectomy (MRM) without delayed reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing neoadjuvant chemotherapy subsequently subjected to conservative surgery (Quadrantectomy/lumpectomy), Oncoplastic surgery second level or conservative mastectomy with breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Development of a new scoring system | 2016-2021
  Definition of a scoring system aimed to perform the radicality desease and aesthetic outcomes in line with expectance of patients

SECONDARY OUTCOMES:
Evaluation of outcome disease | 2016-2021
  Capacity of the new score system to avoid loco-regional disease; Distant disease and Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Franceschini, Prof., Principal Investigator — IRCCS Policlinico Agostino Gemelli - Roma

IPD SHARING:
Plan to Share IPD: Undecided